CLINICAL TRIAL: NCT01032837
Title: A Randomized, Multicenter Trial of Oseltamivir [Tamiflu] Doses of 75 mg for 5 or 10 Days Versus 150 mg for 5 or 10 Days to Evaluate the Effect on the Duration of Viral Shedding in Influenza Patients With Pandemic (H1N1) 2009
Brief Title: A Study of Tamiflu (Oseltamivir) for Treatment of Influenza With a Focus on (H1N1) 2009 Flu Strain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study closed prematurely due to the end of the influenza (H1N1) 2009 pandemic
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV22155
Record Dates: First submitted 2009-12-10; First posted 2009-12-16 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Oseltamivir standard dose 5 days (Experimental): Adults and children 13 years and older received 75 mg oseltamivir and a placebo capsule twice daily for 5 days. Children aged 1 - 12 years received a weight-based dose (from 30 to 75 mg) oseltamivir suspension and placebo suspension orally twice daily for 5 days. Participants received matching placebo for the second 5 days of treatment.
  Interventions: Drug: Oseltamivir; Drug: Placebo
- Oseltamivir standard dose 10 days (Experimental): Adults and children 13 years and older received 75 mg oseltamivir and a placebo capsule twice daily for 10 days. Children aged 1 - 12 years received a weight-based dose (from 30 to 75 mg) oseltamivir suspension and placebo suspension orally twice daily for 10 days.
  Interventions: Drug: Oseltamivir; Drug: Placebo
- Oseltamivir high dose 5 days (Experimental): Adults and children 13 years and older received 150 mg (2 x 75 mg) oseltamivir capsules twice daily for 5 days. Children aged 1 - 12 years received a weight-based dose (from 60 to 150 mg) oseltamivir suspension orally twice daily for 5 days. Participants received matching placebo for the second 5 days of treatment.
  Interventions: Drug: Oseltamivir; Drug: Placebo
- Oseltamivir high dose 10 days (Experimental): Adults and children 13 years and older received 150 mg (2 x 75 mg) oseltamivir capsules twice daily for 10 days. Children aged 1- 12 years received a weight-based dose (from 60 to 150 mg) oseltamivir suspension orally twice daily for 10 days.
  Interventions: Drug: Oseltamivir; Drug: Placebo

INTERVENTIONS:
Drug: Oseltamivir — Oseltamivir capsules for participants ≥ 13 years.
  Other Names: Tamiflu
Drug: Oseltamivir — Pediatric suspension for participants aged ≤ 12 years.
  Other Names: Tamiflu
Drug: Placebo — Matching placebo provided as capsules and as a suspension.

SUMMARY:
This randomized, double-blind, multi-center study of Tamiflu (Oseltamivir) will evaluate the efficacy against viral activity, the effectiveness in resolving the disease symptoms, and the safety and tolerability in patients with influenza. Patients with (H1N1) 2009 influenza strain or influenza A are eligible for this study. Patients will be randomized to one of four treatment regimens. Patients will receive oral doses of either 75 mg (adults) or 150 mg (adults) of study drug twice daily for 5 or 10 consecutive days. The dose will be body weight-adjusted for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric, adolescent and adult patients >/=1 year of age
* Fever >/=37.8 degrees C or at least one respiratory symptom (cough, coryza, sore throat, or rhinitis)
* Positive rapid diagnostic test for pandemic (H1N1) 2009 virus or influenza A in the 24 hours prior to the first dose of study drug
* </=96 hours between onset of influenza-like illness and first dose of oseltamivir

Exclusion Criteria:

* Currently receiving any form of renal replacement therapy including hemodialysis, peritoneal dialysis, or hemofiltration
* History of chronic renal failure or clinical suspicion of renal failure at baseline
* Clinical evidence of hepatic compensation at the time of randomization
* Known HIV infection
* Vaccination with live attenuated influenza vaccine (LAIV) in the two weeks prior to first dose of study medication

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (94):
- United States (94):
  - Tuscaloosa, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Jonesboro, Arkansas
  - Carmichael, California
  - Downey, California
  - Fountain Valley, California
  - Huntington Beach, California
  - Lomita, California
  - National City, California
  - Paramount, California
  - Sacramento, California
  - San Diego, California
  - Colorado Springs, Colorado
  - DeLand, Florida
  - Fleming Island, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Largo, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Saint Cloud, Florida
  - Atlanta, Georgia
  - Idaho Falls, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Dubuque, Iowa
  - Overland Park, Kansas
  - Bardstown, Kentucky
  - Madisonville, Kentucky
  - Lake Charles, Louisiana
  - Mandeville, Louisiana
  - Meltairie, Louisiana
  - Shreveprt, Louisiana
  - Brockton, Massachusetts
  - Stevensville, Michigan
  - Bridgeton, Missouri
  - St Louis, Missouri
  - Bozeman, Montana
  - Bellevue, Nebraska
  - Freemont, Nebraska
  - Haddon Heights, New Jersey
  - Sicklerville, New Jersey
  - Camillus, New York
  - Endwell, New York
  - Johnson City, New York
  - Asheboro, North Carolina
  - Burlington, North Carolina
  - Greensboro, North Carolina
  - Harrisburg, North Carolina
  - Mooresville, North Carolina
  - Morganton, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Bismarck, North Dakota
  - Canal Fulton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Ashland, Oregon
  - Medford, Oregon
  - Collegeville, Pennsylvania
  - Erie, Pennsylvania
  - Jefferson Hills, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Reading, Pennsylvania
  - Scotland, Pennsylvania
  - Upland, Pennsylvania
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - Bedford, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - New Braunfels, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Clinton, Utah
  - Magna, Utah
  - Salt Lake City, Utah
  - Saratoga Springs, Utah
  - West Jordan, Utah
  - Richmond, Virginia
  - Vienna, Virginia
  - Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Started | 26 | 26 | 25 | 25
Intent-to-Treat | 26 (All patients randomized who received at least one dose of study medication.) | 26 (All patients randomized who received at least one dose of study medication.) | 25 (All patients randomized who received at least one dose of study medication.) | 24 (All patients randomized who received at least one dose of study medication.)
Completed | 26 (Represents patients who completed treatment.) | 23 (Represents patients who completed treatment.) | 24 (Represents patients who completed treatment.) | 22 (Represents patients who completed treatment.)
Not Completed | 0 | 3 | 1 | 3
Not completed — Adverse event/internal illness | 0 | 1 | 0 | 1
Not completed — Withdrew consent | 0 | 2 | 0 | 1
Not completed — Failed to return | 0 | 0 | 1 | 0
Not completed — Refused treatment | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days | Total
Number analyzed (Participants) | 26 | 26 | 25 | 24 | 101
Age, Customized [Number; unit: participants] — Overall number of baseline participants is based on the Intent-to-Treat population.
  participants
    1 to <13 years | 7 | 7 | 7 | 6 | 27
    13 to ≤18 years | 3 | 2 | 5 | 3 | 13
    >18 years | 16 | 17 | 13 | 15 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 14 | 12 | 54
  Male | 13 | 11 | 11 | 12 | 47
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 2 | 1 | 0 | 4
  Black | 2 | 1 | 3 | 4 | 10
  White | 23 | 23 | 20 | 20 | 86
  White/Black | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Cessation of Viral Shedding
Description: The time to cessation of viral shedding was measured by viral culture and defined as the time from treatment initiation to the time of the first negative culture with no subsequent positive cultures. Any patient with a positive culture at the last sample time was censored at that time point. Median time to cessation was estimated from the Kaplan-Meier curve.
Time Frame: Day 1 to Day 40
Population: ITT infected (ITTI) Population, including all patients randomized who received at least one dose of study medication with laboratory confirmation of pandemic (H1N1) 2009 influenza infection, excluding patients infected with oseltamivir-resistant influenza A H1N1 H275Y at baseline and patients not shedding virus at baseline.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Number analyzed (Participants) | 19 | 18 | 16 | 17
hours | 65.6 [47.5 to 79.9] | 70.8 [62.1 to 101.7] | 58.1 [27.3 to 93.3] | 74.1 [48.6 to 117.5]

2. Secondary Outcome: Percentage of Participants With Viral Shedding by Clinic Visit as Measured by Viral Culture
Description: Viral shedding was measured by viral culture from samples obtained from nasal and throat swabs and performed by the central laboratory.
Time Frame: Baseline and Days 3, 6, 8, 11, 15 and 40
Population: ITTI
Measure: Number; unit: percentage of participants
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Number analyzed (Participants) | 19 | 18 | 16 | 17
percentage of participants
  Baseline (n=19, 18, 16, 17) | 100 | 100 | 100 | 100
  Day 3 (n=19, 17, 15, 15) | 37 | 61 | 44 | 53
  Day 6 (n=19, 17, 15, 15) | 0 | 0 | 6 | 12
  Day 8 (n=18, 17, 15, 15) | 5 | 0 | 0 | 6
  Day 11 (n=18, 18, 15, 14) | 5 | 11 | 0 | 0
  Day 15 (n=18, 14, 15, 12) | 0 | 0 | 0 | 0
  Day 40 (n=16, 15, 16, 14) | 5 | 11 | 0 | 12

3. Secondary Outcome: Percentage of Participants With Viral Shedding by Clinic Visit as Measured by Reverse Transcriptase Polymerase Chain Reaction
Description: Viral shedding was measured by reverse transcriptase polymerase chain reaction (RT-PCR) from samples obtained from nasal and throat swabs and performed by the central laboratory.
Time Frame: Baseline and Days 3, 6, 8, 11, 15 and 40
Population: ITTI
Measure: Number; unit: percentage of participants
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Number analyzed (Participants) | 19 | 18 | 16 | 17
percentage of participants
  Baseline (n=19, 18, 16, 17) | 89 | 100 | 100 | 100
  Day 3 (n=19, 17, 15, 15) | 79 | 83 | 69 | 76
  Day 6 (n=19, 17, 16, 15) | 26 | 28 | 50 | 47
  Day 8 (n=18, 17, 15, 15) | 11 | 11 | 13 | 12
  Day 11 (n=18, 18, 15, 14) | 5 | 6 | 25 | 18
  Day 15 (n=18, 14, 15, 12) | 0 | 6 | 0 | 6
  Day 40 (n=16, 15, 16, 14) | 5 | 6 | 6 | 0

4. Secondary Outcome: Change From Baseline in Influenza Titer Measured by Viral Culture
Description: Influenza virus titer measured by viral culture and expressed on a Log10 scale of the 50% Tissue Culture Infective Dose (TCID50; amount of virus required to kill 50% of inoculated tissue culture cells).
Time Frame: Baseline, Days 2 through 15
Population: ITTI
Measure: Mean (Standard Deviation); unit: Log10 TCID50
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Number analyzed (Participants) | 19 | 18 | 16 | 17
Log10 TCID50
  Baseline (n=19, 18, 16, 17) | 3.74 (1.478) | 4.06 (1.235) | 4.14 (1.338) | 4.54 (0.746)
  Day 2 (n=19, 18, 15, 17) | -1.82 (1.457) | -1.17 (1.138) | -1.97 (1.584) | -1.15 (1.425)
  Day 3 (n=19, 18, 15, 17) | -2.38 (1.670) | -2.18 (1.221) | -2.95 (1.286) | -2.88 (1.296)
  Day 4 (n=19, 18, 15, 17) | -3.18 (1.511) | -3.29 (1.129) | -3.33 (1.368) | -3.76 (0.859)
  Day 5 (n=19, 18, 16, 17) | -3.00 (1.656) | -3.43 (1.140) | -3.45 (1.453) | -3.91 (0.765)
  Day 6 (n=19, 18, 15, 17) | -3.22 (1.488) | -3.56 (1.235) | -3.45 (1.530) | -3.99 (0.726)
  Day 7 (n=19, 18, 16, 17) | -3.22 (1.469) | -3.53 (1.218) | -3.58 (1.331) | -4.04 (0.746)
  Day 8 (n=19, 18, 15, 17) | -3.18 (1.457) | -3.56 (1.235) | -3.65 (1.385) | -4.04 (0.746)
  Day 9 (n=19, 18, 14, 16) | -3.24 (1.478) | -3.53 (1.218) | -3.57 (1.381) | -4.08 (0.688)
  Day 10 (n=19, 18, 15, 16) | -3.21 (1.463) | -3.50 (1.260) | -3.55 (1.334) | -4.14 (0.652)
  Day 11 (n=19, 16, 16, 15) | -3.22 (1.469) | -3.42 (1.524) | -3.64 (1.338) | -4.08 (0.632)
  Day 12 (n=19, 18, 15, 15) | -3.11 (1.669) | -3.47 (1.289) | -3.63 (1.385) | -4.10 (0.653)
  Day 13 (n=19, 18, 16, 15) | -3.17 (1.458) | -3.43 (1.248) | -3.64 (1.338) | -4.10 (0.653)
  Day 14 (n=18, 18, 15, 15) | -3.17 (1.488) | -3.56 (1.235) | -3.55 (1.334) | -4.10 (0.653)
  Day 15 (n=18, 17, 14, 15) | -3.14 (1.456) | -3.50 (1.250) | -3.55 (1.401) | -4.10 (0.653)

5. Secondary Outcome: Number of Participants With Development of Oseltamivir-Resistant Influenza Virus
Description: The last positive viral isolate from each patient was tested for reduced sensitivity to oseltamivir. Phenotypic assay was performed to determine the susceptibility of the last positive viral isolate from each patient. If required, a genotypic assay to determine the contribution of both the neuraminidase (NA) and hemagglutinin (HA) genes to decreased susceptibility was also performed.
Time Frame: 40 days
Population: ITTI Population
Measure: Number; unit: participants
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Number analyzed (Participants) | 19 | 18 | 16 | 17
participants | 0 | 1 | 1 | 0

6. Secondary Outcome: Time to Resolution of Fever
Description: Temperature was recorded by the patient in a diary twice daily for 10 days and once daily thereafter. Fever was defined as a body temperature greater than or including 37.8 degrees Celsius (or ≥ 100.04 Fahrenheit). Time to resolution of fever was defined as the total number of hours from the first dose of study medication to the first time at which temperature is ≤ 37.2 degrees Celsius and lasts at least 21.5 hours. Patients who were still febrile at the end of the study period were censored at that time.
Time Frame: Day 1 through Day 40
Population: ITTI population with fever at Baseline.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Number analyzed (Participants) | 10 | 6 | 8 | 3
hours | 19.3 [10.6 to 58.4] | 35.5 [12.7 to 53.1] | 24.9 [15.7 to 45.2] | 20.0 [15.9 to 74.3]

7. Secondary Outcome: Time to Alleviation of All Clinical Symptoms - Children
Description: Daily influenza-like symptoms (such as poor appetite, irritability, low energy, nasal congestion, runny nose etc) were recorded in a diary on a scale from 0 (no problem) to 3 (major problem). A patient is considered free of all clinical influenza symptoms if all symptoms were checked as 'no problem' or 'minor problem' (i.e., symptom score ≤1). Time to alleviation of all clinical symptoms was defined as the number of hours from the first dose to the first time the patient had alleviation of all symptoms. Patients without alleviation of symptoms were censored at the last available assessment.
Time Frame: Day 1 to Day 40
Population: ITTI population including children only (ages 1 - 12 years).
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Number analyzed (Participants) | 6 | 4 | 4 | 3
hours | 176.8 [67.5 to 302.0] | 127.7 [32.6 to 281.8] | 118.8 [46.3 to 228.2] | 123.1 [7.1 to 232.3]

8. Secondary Outcome: Time to Alleviation of All Clinical Symptoms - Adults
Description: Daily influenza-like symptoms (such as nasal congestion, sore throat, cough, aches and pains, fatigue, headache, chills) were recorded in a diary on a scale from 0 (absent) to 3 (severe). A patient is considered free of all clinical influenza symptoms if all symptoms were checked as 'absent' or 'mild' (i.e., symptom score ≤1). Time to alleviation of all clinical symptoms was defined as the number of hours from the first dose to the first time the patient had alleviation of all symptoms. Patients without alleviation of symptoms were censored at the last available assessment.
Time Frame: Day 1 to Day 40
Population: ITTI population including adults only (>12 years old).
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Number analyzed (Participants) | 13 | 14 | 12 | 14
hours | 140.0 [99.8 to 183.1] | 181.8 [87.0 to 354.6] | 146.8 [109.1 to 237.8] | 94.9 [57.2 to 261.2]

9. Secondary Outcome: Number of Participants Who Developed Secondary Illnesses During the Study
Description: The number of participants who developed secondary illnesses due to influenza, including four pre-defined adverse events: otitis media, bronchitis, pneumonia, or sinusitis at any time during the study.
Time Frame: Day 1 through Day 40
Population: ITTI population
Measure: Number; unit: participants
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Number analyzed (Participants) | 19 | 18 | 16 | 17
participants
  Bronchitis | 1 | 0 | 0 | 0
  Otitis media | 0 | 0 | 0 | 0
  Pneumonia | 0 | 0 | 0 | 0
  Sinusitis | 0 | 0 | 0 | 2
  Any secondary illness | 1 | 0 | 0 | 2

10. Secondary Outcome: Number of Participants Who Developed Secondary Illnesses That Were Treated With Antibiotics
Description: The number of participants who developed secondary illnesses due to influenza, including otitis media, bronchitis, pneumonia, or sinusitis at any time during the study which were treated with antibiotics.
Time Frame: Day 1 through Day 40
Population: ITTI population
Measure: Number; unit: participants
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Number analyzed (Participants) | 19 | 18 | 16 | 17
participants | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Arm/Group | Oseltamivir Standard Dose 5 Days | Oseltamivir Standard Dose 10 Days | Oseltamivir High Dose 5 Days | Oseltamivir High Dose 10 Days
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 3/26 | 5/26 | 3/25 | 6/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir Standard Dose 5 Days (N=26) | Oseltamivir Standard Dose 10 Days (N=26) | Oseltamivir High Dose 5 Days (N=25) | Oseltamivir High Dose 10 Days (N=24)
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 6
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.